CLINICAL TRIAL: NCT05128448
Title: Comparative Effects of Two Procedures for the Management of Posterior Shoulder Tightness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Rafael Baeske, Principal investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FACCAT
Record Dates: First submitted 2021-10-17; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Posterior Shoulder Tightness
MeSH Terms: interventions — Movement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All measurements will be conducted by research assistants unaware of the interventions applied. Statistical analyses will be performed by a blinded research assistant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilisation with movement (MWM) (Experimental): With the participant standing, the restricted shoulder will rest on the clinician's shoulder in the following starting position: 90 degrees of glenohumeral abduction and 90 degrees of elbow flexion and hand holding a treatment belt. The belt will loop around the clinician and patient and will be held by the participant's contralateral hand. The clinician will apply and sustain a pain free caudal or posterolateralcaudal humeral head mobilisation force (whichever is more comfortable to the subject), followed by an active internal rotation (IR) performed by the patient. The IR movement will be performed to a pain free end of range. If possible, an overpressure with be requested, this is achieved by pulling the belt with the contralateral hand. The overpressure should not produce pain, if it does, it will not be performed.
  3 sets of 8 repetitions will be applied, sustaining the end of available range for 2 seconds. An interval of 45 seconds will be respected amongst the repetitions.
  Interventions: Other: Mobilisation with movement (MWM)
- Cross-body stretch (Active Comparator): With the participant standing, the restricted shoulder will be self-stretched by conducting a horizontal adduction in 90 degrees of shoulder flexion to a level tolerated by the participant. This position will be held for thirty seconds and repeated four times. An interval of forty five seconds will be respected amongst the repetitions.
  Interventions: Other: Cross-body stretch (CBS)

INTERVENTIONS:
Other: Cross-body stretch (CBS) — CBS is a self administered stretch that aims to stretch posterior shoulder structures
  Arms: Cross-body stretch
Other: Mobilisation with movement (MWM) — WMW is a musculoskeletal procedure that aims to improve restricted and/or painful range of movement
  Arms: Mobilisation with movement (MWM)

SUMMARY:
This study aims to compare the effects of a self-stretch procedures versus a clinician applied musculoskeletal procedure in individuals with posterior shoulder tightness.

DETAILED DESCRIPTION:
Posterior shoulder mobility has been considered a contributing factor to shoulder related movement dysfunction. There is evidence indicating that posterior shoulder tightness (PST) might be present in individuals with impingement related symptoms, post-operative conditions and overhead athletes. Several studies have investigated the effects of musculoskeletal procedures (joint mobilisations and stretch) in subjects with posterior shoulder tightness (PST). This cross-over design aims to compare the differences between a well-established procedure - the crossbody stretch - versus mobilisation with movement, on range of motion and pain pressure threshold of asymptomatic individuals with unilateral PST.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic individuals without any history of shoulder pain necessitating medical attention.
* Presence of unilateral restriction of at least 10 degrees of internal rotation deficit during the internal rotation mobility test in 90 degrees of shoulder abduction.

Exclusion Criteria:

* Asymptomatic individuals that present with shoulder pain on the assessment day.
* Individuals with chronic conditions not affecting the shoulder.
* Individuals with clinical depression.
* Individuals that used analgesic and/or anti-inflammatory medication in the previous 24 hours of assessment.
* Individuals with fibromialgia.
* Individuals engaged in overhead sports.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-10-17 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Horizontal adduction | change immediately after the intervention
  Horizontal adduction in 90 degrees of shoulder flexion
Internal rotation | change immediately after the intervention
  Internal rotation at 90 degrees of shoulder abduction

SECONDARY OUTCOMES:
Mechanical sensitivity | change immediately after the intervention
  Pain pressure threshold with an algometer (Wagner instruments, FPX 25)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Faria Silva, PhD, Study Chair — Federal University of Health Science of Porto Alegre
Locations (1):
- Faculdades Integradas de Taquara, Taquara, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Data will be provided on reasonable request.

REFERENCES:
- [Background] Picavet HS, Schouten JS. Musculoskeletal pain in the Netherlands: prevalences, consequences and risk groups, the DMC(3)-study. Pain. 2003 Mar;102(1-2):167-78. doi: 10.1016/s0304-3959(02)00372-x. PMID 12620608
- [Background] Hall K, Borstad JD. Posterior Shoulder Tightness: To Treat or Not to Treat? J Orthop Sports Phys Ther. 2018 Mar;48(3):133-136. doi: 10.2519/jospt.2018.0605. PMID 29490601
- [Background] Schwartz C, Croisier JL, Bruls O, Denoel V, Forthomme B. Tight shoulders: A clinical, kinematic and strength comparison of symptomatic and asymptomatic male overhead athletes before and after stretching. Eur J Sport Sci. 2021 May;21(5):781-791. doi: 10.1080/17461391.2020.1785015. Epub 2020 Jul 7. PMID 32635824
- [Background] Rosa DP, Borstad JD, Ferreira JK, Camargo PR. The Influence of Glenohumeral Joint Posterior Capsule Tightness and Impingement Symptoms on Shoulder Impairments and Kinematics. Phys Ther. 2019 Jul 1;99(7):870-881. doi: 10.1093/ptj/pzz052. PMID 30921461
- [Background] Tyler TF, Nicholas SJ, Lee SJ, Mullaney M, McHugh MP. Correction of posterior shoulder tightness is associated with symptom resolution in patients with internal impingement. Am J Sports Med. 2010 Jan;38(1):114-9. doi: 10.1177/0363546509346050. Epub 2009 Dec 4. PMID 19966099
- [Background] Salamh PA, Kolber MJ, Hegedus EJ, Cook CE. The efficacy of stretching exercises to reduce posterior shoulder tightness acutely in the postoperative population: a single blinded randomized controlled trial. Physiother Theory Pract. 2018 Feb;34(2):111-120. doi: 10.1080/09593985.2017.1376020. Epub 2017 Sep 13. PMID 28901811
- [Background] Salamh PA, Liu X, Kolber MJ, Hanney WJ, Hegedus EJ. The reliability, validity, and methodologic quality of measurements used to quantify posterior shoulder tightness: a systematic review of the literature with meta-analysis. J Shoulder Elbow Surg. 2019 Jan;28(1):178-185. doi: 10.1016/j.jse.2018.07.013. Epub 2018 Oct 1. PMID 30287146
- [Background] Mine K, Nakayama T, Milanese S, Grimmer K. Effectiveness of Stretching on Posterior Shoulder Tightness and Glenohumeral Internal-Rotation Deficit: A Systematic Review of Randomized Controlled Trials. J Sport Rehabil. 2017 Jul;26(4):294-305. doi: 10.1123/jsr.2015-0172. Epub 2016 Aug 24. PMID 27632891
- [Background] Salamh PA, Liu X, Hanney WJ, Sprague PA, Kolber MJ. The efficacy and fidelity of clinical interventions used to reduce posterior shoulder tightness: a systematic review with meta-analysis. J Shoulder Elbow Surg. 2019 Jun;28(6):1204-1213. doi: 10.1016/j.jse.2018.12.006. Epub 2019 Mar 20. PMID 30902594
- [Background] Kang MH, Oh JS. Effects of self-stretching with mobilization on shoulder range of motion in individuals with glenohumeral internal rotation deficits: a randomized controlled trial. J Shoulder Elbow Surg. 2020 Jan;29(1):36-43. doi: 10.1016/j.jse.2019.08.007. Epub 2019 Oct 15. PMID 31627965
- [Background] Hall K, Lewis J, Moore A, Ridehalgh C. Posterior shoulder tightness; an intersession reliability study of 3 clinical tests. Arch Physiother. 2020 Jul 29;10:14. doi: 10.1186/s40945-020-00084-w. eCollection 2020. PMID 32742721
- [Result] Oliveira VMA, Pitangui ACR, Gomes MRA, Silva HAD, Passos MHPD, Araujo RC. Shoulder pain in adolescent athletes: prevalence, associated factors and its influence on upper limb function. Braz J Phys Ther. 2017 Mar-Apr;21(2):107-113. doi: 10.1016/j.bjpt.2017.03.005. Epub 2017 Mar 17. PMID 28460708